CLINICAL TRIAL: NCT05194579
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, 2-WAY CROSSOVER STUDY ASSESSING PHARMACOKINETIC COMPARABILITY OF TWO PF-06881894 PRESENTATIONS, ON-BODY INJECTOR AND PREFILLED SYRINGE, IN HEALTHY PARTICIPANTS
Brief Title: Pharmacokinetic Comparability Study in Healthy Participants - PF-06881894 On-Body Injector Relative to Prefilled Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C1221007; OBI (Other: Alias Study Number)
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: on-body injector; OBI; febrile neutropenia; pegfilgrastim
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06881894 by on-body injector (OBI) (Other): PF-06881894 given by on-body injector (OBI) as test arm, 6 mg administered as a single SC injection
  Interventions: Combination Product: PF-06881894 by on-body injector
- PF-06881894 by prefilled syringe (PFS) (Other): PF-06881894 given by prefilled syringe (PFS) as reference arm, 6 mg administered as a single SC injection
  Interventions: Combination Product: PF-06881894 by prefilled syringe

INTERVENTIONS:
Combination Product: PF-06881894 by on-body injector — PF-06881894 given by on-body injector (OBI), 6 mg administered as a single SC injection
  Other Names: on-body injector
  Arms: PF-06881894 by on-body injector (OBI)
Combination Product: PF-06881894 by prefilled syringe — PF-06881894 given by prefilled syringe (PFS), 6 mg administered as a single SC injection
  Arms: PF-06881894 by prefilled syringe (PFS)

SUMMARY:
This will be an open-label, randomized, 2-treatment, 2-period, crossover single-dose study in approximately 134 healthy adult participants. Participants will be randomized into 2 sequences of treatment as described in the following table of Intervention Groups and Duration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants who, at the time of screening, are between the ages of 18 and 65 years, inclusive.
* Participants will include healthy individuals, with healthy being defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including BP and PR measurement, 12-lead ECG, chest X-ray, or clinical laboratory tests.
* Participants agree to abstain from the use of tobacco- or nicotine-containing products for at least 90 days prior to dosing and have a negative urine screen for cotinine at Screening.
* Participants agree to abstain from alcohol consumption for at least 48 hours prior to Day 1 of dosing in each study period and have a negative screen for alcohol.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI between 19 and 30 kg/m2, inclusive, and body weight of not<50 kg or >100 kg.
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, injuries to subcutaneous tissue at the injection site).
* Any clinically significant, as determined by the investigator, abnormal laboratory evaluations, including HIVAb, HBVsAg, HBVcAb, HCVAb and liver function taken at Screening. The negative HIVAb status will be confirmed at Screening, and all HIV results will be maintained confidentially by the study site.
* History of malignancy, including current malignancy, with the exception of adequately treated squamous or basal cell carcinoma of the skin or cervical carcinoma in situ within 5 years.
* Surgery within the 4 months prior to Screening.
* History of splenic rupture (or participant who is asplenic), pulmonary infiltrate or pneumonia, sickle cell disease, chronic neutropenia, thrombocytopenia, or vasculitis.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of biological growth factor exposure, including but not limited to pegfilgrastim, filgrastim and other G-CSFs in the context of treatment, prophylaxis, peripheral blood stem cell mobilization, or previous investigational study setting. This also includes exclusion for history of interferon, epoetin, and IVIG exposure.
* Receipt of live vaccination, or exposure to communicable viral diseases such as chicken pox, varicella, mumps, measles, or COVID-19 within the 4 weeks prior to Screening.
* Use of any prescription medicine (with the exception of contraceptives) within 7 days or at least 5 half-lives, whichever was longer. Use of oral or parenteral anticoagulant or antiplatelet agents and corticosteroids should be specifically queried.
* Administration of a drug by depot injection (with the exception of depot contraception) within 30 days prior to the initial study drug administration or 5 half-lives of that drug, whichever is longer.
* Use of over the counter medications, including aspirin and non-steroidal anti-inflammatory drugs, or natural preparations (dietary supplement or herbal product) within 7 days of the first dose of PF-06881894 or at least 5 half-lives, whichever is longer. Vitamins and calcium supplements are allowed (not to exceed 100% Daily Value). As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of non-prescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Females using post-menopausal hormone replacement therapy may be eligible to participate in this study if they are willing to discontinue therapy at least 28 days prior to the first dose of study treatment and remain off hormonal therapy for the duration of the study. Hormonal contraceptives that meet the requirements of this study are allowed to be used in participants who are women of childbearing potential.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention (whichever is longer) prior to study entry and/or during study participation. If a participant receives a vaccine or other medical product for the prevention or treatment of COVID-19 authorized under an Emergency Use Authorization, this would not be considered an investigational medical product.
* Hematologic laboratory abnormalities at screening or the Day -5 to Day -4 visit including leukocytosis (defined as total leukocytes >11,000/μL), leukopenia (defined as total leukocytes <4000/μL), neutropenia (defined as ANC <1500/μL) or thrombocytopenia (defined as platelet count of <150,000/μL).
* A positive urine drug test.
* A positive SARS-CoV-2 infection determined by PCR at screening or Day -5 to Day -4, or determined by a positive COVID-19 antigen test (if performed as part of an investigator site policy).
* Screening supine BP >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Screening supine 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the participant's eligibility.
* Participants with the following abnormalities in clinical laboratory tests at screening or the Day -5 to Day -4 visit, as assessed by the study specific laboratory will be confirmed by a single repeat test, if deemed necessary. Then the investigator (in consultation with the medical monitor) will determine if the laboratory abnormality is clinically significant and sufficient to exclude the participant from the study.

Lack of adequate hepatic reserve, defined by AST/SGOT or ALT/SGPT >= 1.5 × ULN of the reference laboratory; TBili >= 1.5 × ULN; participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is <= ULN.

Lack of renal reserve, defined by serum creatinine of >= 1.2 × ULN for reference laboratory or eGFR of <= 80 mL/minute; or known history of glomerulonephritis.

* Drug sensitivity, allergic reaction to, or known hypersensitivity/idiosyncratic reaction to E coli -derived proteins, pegfilgrastim, filgrastim, other G-CSFs or any component of the product or known hypersensitivity to pegylated products or acrylic adhesives. Participants with the rare heredity problem of fructose intolerance are excluded due to the excipient sorbitol.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Pregnant female participants, breastfeeding female participants, and male participants able to father children and female participants of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of study intervention.
* Blood donation (including plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing OR had a transfusion of any blood product within 90 days prior to Screening.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol. Male participants with pregnant partners are not to be enrolled in the study, even if the participant is willing to comply with the contraception lifestyle requirements and use a highly effective method of contraception consistently and correctly for the duration of the study and for at least 28 days after the last dose of study intervention.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Clinical Trials of Texas, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1221007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, randomized, 2-treatment (PF-06881894 via prefilled syringe [PFS] or PF-06881894 via on-body injector [OBI]), 2-period, crossover single-dose study. A total of 371 participants were screened for this study; 141 participants were randomized to treatment and treated.
Groups:
- PF-06881894 PFS=>PF-06881894 OBI: Participants received PF-06881894 administered subcutaneously (SC) via PFS on Day 1 of Period 1, then followed by PF-06881894 administered SC via OBI on Day 1 of Period 2. There was a wash out period of at least 56 days between the 2 treatments.
- PF-06881894 OBI=>PF-06881894 PFS: Participants received PF-06881894 administered SC via OBI on Day 1 of Period 1, then followed by PF-06881894 administered SC via PFS on Day 1 of Period 2. There was a wash out period of at least 56 days between the 2 treatments.
Period: Overall Study
Arm/Group | PF-06881894 PFS=>PF-06881894 OBI | PF-06881894 OBI=>PF-06881894 PFS
Started | 70 | 71
Assigned to Treatment | 70 | 71
Completed | 64 | 63
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Refused further study procedures | 0 | 1
Not completed — Protocol deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized and received at least 1 dose of study intervention (regardless of complete or incomplete dose).
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06881894 PFS=>PF-06881894 OBI | PF-06881894 OBI=>PF-06881894 PFS | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (13.09) | 40.2 (11.68) | 39.7 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 36 | 43 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 42 | 82
  Not Hispanic or Latino | 30 | 27 | 57
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 52 | 51 | 103
  Black or African American | 12 | 13 | 25
  Asian | 4 | 5 | 9
  American Indian or Alaska Native | 0 | 1 | 1
  Unknown | 1 | 0 | 1
  Multiracial | 1 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (2.62) | 26.5 (2.47) | 26.3 (2.55)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of PF-06881894
Description: Cmax of PF-06881894 was defined as maximum serum concentration of PF-06881894. Observed directly from data.
Time Frame: Within 1 hour prior to dose (Hour 0) and at 0.167 (10 min), 0.5, 1, 3, 6, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 and 288 hours post-dose
Population: The analysis population for each arm included all randomized participants who were fully dosed and had at least 1 valid pharmacokinetic (PK) primary result in at least 1 treatment period. "Number of Participants Analyzed" signifies number of participants evaluable/non-missing for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- PF-06881894 PFS: Participants received PF-06881894 administered SC via PFS on Day 1 of Period 1 or Period 2.
- PF-06881894 OBI: Participants received PF-06881894 administered SC via OBI on Day 1 of Period 1 or Period 2.
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
Number analyzed (Participants) | 136 | 122
nanogram per milliliter (ng/mL) | 131.2 (151) | 161.1 (126)
Statistical Analysis 1: Comparison: PF-06881894 PFS vs PF-06881894 OBI; The null hypothesis was PF-06881894 OBI was not equivalent to PF-06881894 PFS; Test type: Equivalence — Pharmacokinetic equivalence were assessed by constructing the 90% confidence intervals (CIs) for the GMR (test/reference) for Cmax, AUClast and AUCinf. This table displays Cmax statistical analysis; ANOVA; Ratio of Geometric Mean = 117.06, 90% CI 2-sided [103.07 to 132.93]

2. Primary Outcome: Area Under the Serum Drug Concentration-time Profile From Time 0 to the Last Quantifiable Concentration (AUClast) of PF-06881894
Description: AUClast of PF-06881894 was defined as area under the serum drug concentration-time profile from time 0 to the last quantifiable concentration. Linear/Log trapezoidal method was used.
Time Frame: as for outcome 1
Population: The analysis population for each arm included all randomized participants who were fully dosed and had at least 1 valid PK primary result in at least 1 treatment period. "Number of Participants Analyzed" signifies number of participants evaluable/non-missing for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
Number analyzed (Participants) | 136 | 122
nanogram*hour per milliliter (ng*hr/mL) | 4510 (152) | 5791 (129)
Statistical Analysis 1: Comparison: PF-06881894 PFS vs PF-06881894 OBI; The null hypothesis was PF-06881894 OBI was not equivalent to PF-06881894 PFS; Test type: Equivalence — Pharmacokinetic equivalence were assessed by constructing the 90% CIs for the GMR (test/reference) for Cmax, AUClast and AUCinf. This table displays AUClast statistical analysis; ANOVA; Ratio of Geometric Mean = 122.12, 90% CI 2-sided [107.90 to 138.22]

3. Primary Outcome: Area Under the Serum Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06881894
Description: AUCinf of PF-06881894 was defined as area under the serum concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
Number analyzed (Participants) | 123 | 115
ng*hr/mL | 4869 (128) | 6020 (119)
Statistical Analysis 1: Comparison: PF-06881894 PFS vs PF-06881894 OBI; The null hypothesis was PF-06881894 OBI was not equivalent to PF-06881894 PFS; Test type: Equivalence — Pharmacokinetic equivalence were assessed by constructing the 90% CIs for the GMR (test/reference) for Cmax, AUClast and AUCinf. This table displays AUCinf statistical analysis; ANOVA; Ratio of Geometric Mean = 123.75, 90% CI 2-sided [108.75 to 140.82]

4. Secondary Outcome: Time for Cmax (Tmax) of PF-06881894
Description: Tmax of PF-06881894 was defined as time for Cmax. Observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
Number analyzed (Participants) | 136 | 122
hour | 16.0 [6.00 to 48.1] | 16.0 [3.00 to 72.0]

5. Secondary Outcome: Terminal Serum Elimination Half-life (t½) of PF-06881894
Description: Terminal serum elimination half-life (t½) of PF-06881894 was defined as terminal half-life using Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
Number analyzed (Participants) | 123 | 115
hour | 45.89 (13.683) | 47.42 (14.887)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment-emergent were events between first dose and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to study intervention. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. An AESI was one of scientific and medical concern specific to the sponsor's product or programme. Device related AE was an AE related to the use of an investigational medical device. AEs of ISR and ASR included injection site pain, injection site erythema, application site hemorrhage, application site pain, application site discomfort, application site bruise, and application site erythema.
Time Frame: From the first dose on Day 1 of Period 1 to the Period 2 Day 28 Visit (up to 5 months).
Population: All participants who were randomized and received at least 1 dose of study intervention (regardless of complete or incomplete dose). Here, 'Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
Number analyzed (Participants) | 136 | 136
Participants
  Adverse Event (AE) | 101 | 107
  Serious Adverse Event (SAE) | 0 | 0
  AE of Special Interest (AESI) | 13 | 23
  Device Related AE | 3 | 11
  AE of Injection Site Reaction (ISR) and Application Site Reaction (ASR) | 13 | 23

ADVERSE EVENTS:
Time Frame: From the first dose on Day 1 of Period 1 to the Period 2 Day 28 Visit (up to 5 months).
Description: Adverse events analysis population included all participants who were randomized and received at least 1 dose of study intervention (regardless of complete or incomplete dose).
Arm/Group | PF-06881894 PFS | PF-06881894 OBI
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/136
Other Adverse Events (participants affected / at risk) | 92/136 | 96/136
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06881894 PFS (N=136) | PF-06881894 OBI (N=136)
Nausea (Gastrointestinal disorders) | 9 | 5
Application site erythema (General disorders) | 0 | 13
Injection site pain (General disorders) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 27
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 23
Headache (Nervous system disorders) | 48 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT05194579/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT05194579/SAP_001.pdf